CLINICAL TRIAL: NCT03080727
Title: Intraobserver and Interobserver Reproducibility on Hip Clinical Assessment
Status: Completed | Type: Observational
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Other Study IDs: UFRGS 1.822.689
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Hip Joint

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The functional assessment of the hip joint is complex and challenging. Reproducible measures are necessary to identify changes in the structures and functionality of the hip joint over time and to evaluate the outcomes of treatments. A systematic evaluation process is critical to evidence-based practice. However, there are few studies investigating the reproducibility of these measures such as muscle strength, range of motion (ROM) and hip functionality in healthy subjects.

DETAILED DESCRIPTION:
Twenty subjects were randomized in two different days: (1) First evaluation of muscle strength, range of motion and single-leg squat performed by the evaluator 1; (2) Repeat the first evaluation with 3 different evaluators

ELIGIBILITY:
Inclusion Criteria:

* No complaints of pain or knowledge of hip pathology
* Subjects willing to enroll

Exclusion Criteria:

* Subjects reporting that they can not perform the tests due to pain
* With previous surgery of the hip or pelvis;
* Diabetes Mellitus;
* Neuromuscular or neurological diseases;
* Cardiovascular diseases that prevent the realization of maximum voluntary effort;
* Subjects presenting positive hip clinical tests

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Hip muscle strength | Day 1 (evaluator 1) and after 4 days of rest repeat measures on day 2 with 3 different evaluators
  Measured with isometric hand hel dynamometry

SECONDARY OUTCOMES:
Hip range of motion | Day 1 (evaluator 1) and after 4 days of rest repeat measures on day 2 with 3 different evaluators
  Measured with goniometer

OTHER OUTCOMES:
Single-leg squat | Day 1 (evaluator 1) and after 4 days of rest repeat measures on day 2 with 3 different evaluators
  Hip adduction angle

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil